CLINICAL TRIAL: NCT00022360
Title: An Open-Label Dose-Ranging Study of the Safety of Taurolidine 2% Solution Administered Intravenously to Patients With Recurrent or Progressive High Grade Glioma
Brief Title: Taurolidine in Treating Patients With Recurrent or Progressive Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-01057; CDR0000068808 (Registry Identifier: PDQ (Physician Data Query)); WALLACE-393; NCI-G01-2000
Record Dates: First submitted 2001-08-10; First posted 2004-03-19 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — taurolidine

INTERVENTIONS:
Drug: taurolidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of taurolidine in treating patients who have recurrent or progressive glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of taurolidine in patients with recurrent or progressive high-grade glioma. II. Determine the safety and toxicity of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients. IV. Determine the response in patients treated with this drug.

OUTLINE: This is a dose-escalation study. Patients receive taurolidine IV over 1-4 hours on days 1-5, 8-12, and 15-19. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 1-6 patients receive escalating doses of taurolidine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Patients are followed monthly for 3 months.

PROJECTED ACCRUAL: A total of 4-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma Recurrent or progressive disease after prior cytoreductive surgery, radiotherapy, and adjuvant chemotherapy Ineligible for any additional conventional therapeutic intervention

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: Karnofsky 60-100% Life expectancy: More than 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST/ALT less than 3 times upper limit of normal No indication of acute hepatitis or parenchymal liver disease No significant hepatic disease that would preclude study Renal: Creatinine less than 1.7 mg/dL No significant renal disease that would preclude study Cardiovascular: No significant cardiac disease that would preclude study Other: HIV negative No other active malignancy except curatively treated carcinoma in situ of the cervix or basal cell skin cancer No significant psychiatric disease that would preclude study No significant gastrointestinal disease that would preclude study No known hypersensitivity to taurolidine or its excipients Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior interferon Chemotherapy: See Disease Characteristics At least 2 weeks since prior vincristine At least 3 weeks since prior temozolomide or procarbazine At least 4 weeks since prior nitrosoureas Concurrent polifeprosan 20 with carmustine implant (Gliadel wafers) allowed Endocrine therapy: At least 2 weeks since prior tamoxifen Concurrent corticosteroids allowed Radiotherapy: See Disease Characteristics At least 2 weeks since prior stereotactic radiosurgery Surgery: See Disease Characteristics Other: Recovered from prior therapy At least 30 days since prior investigational drug At least 2 weeks since other prior noncytotoxic agents No other concurrent experimental agent or protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States